CLINICAL TRIAL: NCT02365584
Title: A Phase II, Multicentre, Randomized Controlled Study Evaluating The Quality Of Life In Patients With Inoperable Malignant Bowel Obstruction Treated With Lanreotide Autogel 120 mg in Combination With Standard Care vs. Standard Care Alone (QOL IN IMBO STUDY)
Brief Title: Quality of Life in Patients With Inoperable Malignant Bowel Obstruction
Acronym: QoL in IMBO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to insufficient recruitment.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A-93-52030-279; 2013-003176-12 (EudraCT Number)
Record Dates: First submitted 2015-01-29; First posted 2015-02-19 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Intestinal Obstruction
MeSH Terms: conditions — Intestinal Obstruction | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care and Lanreotide Autogel (Experimental): Standard care according to site clinical practice and Lanreotide Autogel 120 mg by deep subcutaneous route, at the maximal scheduled standard dose of 120 mg/28 days, just for 1 administration.
  Interventions: Drug: lanreotide (Autogel formulation)
- Standard care (No Intervention): Standard care according to site clinical practice.

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — Lanreotide Autogel 120 mg by deep subcutaneous route, at the maximal scheduled standard dose of 120 mg/28 days, just for 1 administration.
  Arms: Standard care and Lanreotide Autogel

SUMMARY:
The primary objective of the study is to evaluate the impact on quality of life of Lanreotide Autogel 120 mg in combination with standard care, in comparison to the standard care alone, in subjects affected by inoperable malignant bowel obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate willingness to participate in the study and to be compliant with any protocol procedure.
* Provision of written informed consent prior to any study related procedure.
* Diagnosis of an inoperable malignant bowel obstruction, confirmed by appropriate imaging report.
* In case of peritoneal carcinomatosis, diagnostic confirmation by CT or MRI scan.
* Confirmed as inoperable after medical advice.
* Patient with a nasogastric tube or presenting with 3 or more episodes of vomiting every day in the last consecutive 48 hours.
* Patient life expectancy must be more than 14 days.

Exclusion Criteria:

* Has operable obstruction or any sub-obstruction.
* Has bowel obstruction due to a non-malignant cause; (hypokaliaemia, drug side-effects, renal insufficiency, etc).
* Has signs of bowel perforation.
* Has prior treatment with somatostatin or any analogue within the previous 60 days.
* Has a known hypersensitivity to any of the study treatments or related compounds.
* Is likely to require treatment during the study with somatostatin or any analogue other than the study treatment.
* Is at risk of pregnancy or lactation, or is likely to father a child during the study. Females of childbearing potential must provide a negative pregnancy test at start of study and must be using oral or double barrier contraception. Non childbearing potential is defined as post-menopause for at least 1 year, surgical sterilisation or hysterectomy at least three months before the start of the study.
* Has any mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (13):
- Italy (13):
  - Ospedale Sacro Cuore di Gesù, U.O.C. Oncologia Medica, Gallipoli, Lecce
  - Ospedali riuniti Ancona- Dipartimento Medicina Interna - Clinica Oncologica, Ancona
  - Centro di Riferimento Oncologico - di Aviano, Dip. di Oncologia Chirurgica- S.O.C. di Chirurgia Oncologica Generale, Aviano
  - Istituto Tumori "Giovanni Paolo II"- Istituto di Ricovero e Cura a Carattere Scientifico, U.O.C. DI ONCOLOGIA MEDICA, Bari
  - Ospedale Sacro Cuore di Gesù - Fatebenefratelli, Benevento
  - Hospice Convento delle Oblate, Florence
  - Azienda Sanitaria Locale n ° 5 "Spezzino" Ospedale Felettino - Oncologia Via del Forno 4, La Spezia
  - I.R.C.C.S. Istituto Scientifico Romagnolo per lo Studio e la cura dei Tumori (I.R.S.T.) srl, Meldola
  - Ospedale San Raffaele IRCCS, Ginecologia oncologica, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori - Struttura Complessa di Cure Palliative, Terapia del Dolore e Riabilitazione, Milan
  - Azienda Ospedaliero - Polo Universitario "Luigi Sacco", Milan
  - A.R.N.A.S. P.O. Civico Benfratelli - Oncologia Medica, Palermo
  - Azienda Ospedaliera Regionale San Carlo- Oncologia Medica, Potenza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to this prospective, randomised, parallel arm, open-label study began on 14 Jan 2015. Patients with a documented diagnosis of inoperable malignant bowel obstruction who had a nasogastric tube (NGT) or presented with ≥ 3 vomiting episodes/day in the last consecutive 48 hours at time of enrolment were recruited to 14 centres in Italy.
Pre-assignment Details: Overall, 43 patients were enrolled and treated in this phase II study. Planned study period duration was 28 days.
Groups:
- Standard Care: Patients received standard care only according to site clinical practice.
- Standard Care + Lanreotide Autogel: Patients received standard care according to site clinical practice and a single administration of Lanreotide Autogel 120 milligrams (mg) by deep subcutaneous injection on Day 1.
Period: Overall Study
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Started | 21 | 22
Completed | 9 | 8
Not Completed | 12 | 14
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease Progression | 9 | 12

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on the intention to treat (ITT) population which included all randomised patients.
Groups:
- Standard Care + Lanreotide Autogel: Patients received standard care according to site clinical practice and a single administration of Lanreotide Autogel 120 mg by deep subcutaneous injection on Day 1.
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel | Total Title
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (9.6) | 62.8 (12.3) | 62.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian / White | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Area Under Curve (AUC) of Edmonton Symptom Assessment System (ESAS) Total Scores Collected for the First 7 Days; Full Analysis Set (FAS)
Description: Quality of Life was assessed using ESAS, evaluating 9 common symptoms in cancer patients: pain, activity, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath. Symptom severity is rated 0-10 on a numerical scale (0=symptom absent; 10=worst severity). ESAS total score is sum of the 9 items (min score=0, max score=90). Low scores indicate good quality of life; high scores indicate strong discomfort. Questionnaire assessments by the patient or by nurse/caregiver in case of patient's physical inability. AUC is area under the line which joins the points defined by plotting ESAS total score on vertical axis and time values on horizontal axis, computed using trapezoidal rule.
  Primary endpoint was analysed using the FAS. LS mean AUC of ESAS total scores during first 7 days is presented.
Time Frame: Baseline (Day 1, before randomisation), Days 2, 3, 4, 5, 6 and 7.
Population: The FAS included all randomised patients who received study therapy, fulfilled the ESAS questionnaire at baseline and had ≥ 5 post-treatment assessments during the first 7 days of the study.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale x time (day)
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 19 | 19
Scores on a scale x time (day) | 179 (12.4) | 190 (12.4)
Statistical Analysis 1: Comparison: Standard Care vs Standard Care + Lanreotide Autogel; Analysis of covariance (ANCOVA), where the AUC was the dependent and the independent was the baseline ESAS total score; Test type: Superiority — The assumptions required for the analysis of covariance (ANCOVA) were to be tested as follows: * The equality of variances was to verified using the Levene's test. If it was significant AUC values were to be properly transformed. * The linear relationship of AUC with the basal total score within treatment group was to be tested by a regression analysis. * The parallelism of the regression lines between groups and the slope non zero value with the appropriate F tests; p = 0.5396, ANCOVA; Adjusted LS Mean Difference = -11, 95% CI 2-sided [-47 to 25], Standard Error of Mean 17.7

2. Secondary Outcome: Mean Change From Baseline in ESAS Total Score; FAS
Description: Quality of Life was assessed using ESAS, evaluating 9 common symptoms in cancer patients: pain, activity, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath. Symptom severity is rated 0-10 on a numerical scale (0=symptom absent; 10=worst severity). ESAS total score is sum of the 9 items (min score=0, max score=90). Low scores indicate good quality of life; high scores indicate strong discomfort. Questionnaire assessments by the patient or by nurse/caregiver in case of patient's physical inability.
  Secondary endpoints were analysed using the ITT population but to permit following the FAS which was used for primary endpoint analysis, ESAS total score results are reported for both the ITT and the FAS. Mean change from baseline of ESAS total score at Days 7, 14 and 28 is presented here for the FAS; a positive change indicates a worsening condition.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: The FAS included all randomised patients who received study therapy, fulfilled the ESAS questionnaire at baseline and had ≥ 5 post-treatment assessments during the first 7 days of the study. Only patients with data available for analysis at each time point are presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 19 | 19
Scores on a scale
  Change at Day 7: number analyzed (Participants) | 18 | 19
  Change at Day 7 | -5.1 (15.7) | 1.9 (18.4)
  Change at Day 14: number analyzed (Participants) | 16 | 14
  Change at Day 14 | -1.3 (21.4) | -7.3 (16.7)
  Change at Day 28: number analyzed (Participants) | 8 | 8
  Change at Day 28 | -6.8 (15.2) | -10.3 (16.7)

3. Secondary Outcome: Mean Change From Baseline in ESAS Total Score; ITT Population
Description: Quality of Life was assessed using ESAS, evaluating 9 common symptoms in cancer patients: pain, activity, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath. Symptom severity is rated 0-10 on a numerical scale (0=symptom absent; 10=worst severity). ESAS total score is sum of the 9 items (min score=0, max score=90). Low scores indicate good quality of life; high scores indicate strong discomfort. Questionnaire assessments by the patient or by nurse/caregiver in case of patient's physical inability.
  Secondary endpoints were analysed using the ITT population but to permit following the FAS which was used for primary endpoint analysis, ESAS total score results are reported for both the ITT and the FAS. Mean change from baseline of ESAS total score at Days 7, 14 and 28 is presented here for the ITT population; a positive change indicates a worsening condition.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: The ITT population included all randomised patients. Only patients with data available for analysis at each time point are presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Scores on a scale
  Change at Day 7: number analyzed (Participants) | 18 | 20
  Change at Day 7 | -5.1 (15.7) | 1.5 (18.1)
  Change at Day 14: number analyzed (Participants) | 16 | 14
  Change at Day 14 | -1.3 (21.4) | -7.3 (16.7)
  Change at Day 28: number analyzed (Participants) | 8 | 8
  Change at Day 28 | -6.8 (15.2) | -10.3 (16.7)

4. Secondary Outcome: Mean Change From Baseline in Single ESAS Items Symptom Scores; ITT Population
Description: Quality of Life was assessed using ESAS, evaluating 9 common symptoms in cancer patients: pain, activity, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath. Symptom severity is rated 0-10 on a numerical scale (0=symptom absent; 10=worst severity). Low scores indicate good quality of life; high scores indicate strong discomfort. Questionnaire assessments by the patient or by nurse/caregiver in case of patient's physical inability.
  Mean change from baseline of each individual ESAS item score at Days 7, 14 and 28 is presented; a positive change indicates a worsening condition.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Scores on a scale
  Change at Day 7: Pain: number analyzed (Participants) | 18 | 20
  Change at Day 7: Pain | -1.8 (3.6) | 0.1 (3.4)
  Change at Day 14: Pain: number analyzed (Participants) | 16 | 13
  Change at Day 14: Pain | -1.3 (3.6) | -1.9 (2.9)
  Change at Day 28: Pain: number analyzed (Participants) | 7 | 6
  Change at Day 28: Pain | -3.0 (3.1) | -1.3 (4.2)
  Change at Day 7: Activity: number analyzed (Participants) | 18 | 20
  Change at Day 7: Activity | -0.3 (2.6) | 0.7 (2.6)
  Change at Day 14: Activity: number analyzed (Participants) | 16 | 13
  Change at Day 14: Activity | -0.3 (3.3) | -0.7 (3.0)
  Change at Day 28: Activity: number analyzed (Participants) | 7 | 6
  Change at Day 28: Activity | -1.4 (2.8) | -0.3 (3.2)
  Change at Day 7: Nausea: number analyzed (Participants) | 18 | 20
  Change at Day 7: Nausea | 0.5 (3.2) | 0.9 (3.2)
  Change at Day 14: Nausea: number analyzed (Participants) | 16 | 13
  Change at Day 14: Nausea | 0.1 (3.8) | 0.5 (4.1)
  Change at Day 28: Nausea: number analyzed (Participants) | 7 | 6
  Change at Day 28: Nausea | -0.6 (4.6) | 0.0 (3.9)
  Change at Day 7: Depression: number analyzed (Participants) | 18 | 20
  Change at Day 7: Depression | -1.8 (3.5) | -1.1 (3.7)
  Change at Day 14 Depression: number analyzed (Participants) | 16 | 13
  Change at Day 14 Depression | -1.9 (3.5) | -2.4 (3.2)
  Change at Day 28: Depression: number analyzed (Participants) | 7 | 6
  Change at Day 28: Depression | -2.6 (1.9) | -3.7 (4.0)
  Change at Day 7: Anxiety: number analyzed (Participants) | 18 | 20
  Change at Day 7: Anxiety | 0.0 (2.7) | -0.2 (3.2)
  Change at Day 14: Anxiety: number analyzed (Participants) | 16 | 13
  Change at Day 14: Anxiety | 0.4 (3.3) | -2.7 (3.8)
  Change at Day 28: Anxiety: number analyzed (Participants) | 7 | 6
  Change at Day 28: Anxiety | -1.1 (1.9) | -1.5 (1.0)
  Change at Day 7: Drowsiness: number analyzed (Participants) | 18 | 20
  Change at Day 7: Drowsiness | -0.7 (2.7) | 0.4 (3.1)
  Change at Day 14: Drowsiness: number analyzed (Participants) | 16 | 13
  Change at Day 14: Drowsiness | -0.1 (3.5) | -0.6 (2.6)
  Change at Day 28: Drowsiness: number analyzed (Participants) | 7 | 6
  Change at Day 28: Drowsiness | -1.9 (3.1) | -1.5 (1.5)
  Change at Day 7: Appetite: number analyzed (Participants) | 18 | 20
  Change at Day 7: Appetite | -0.2 (3.1) | 0.5 (3.2)
  Change at Day 14: Appetite: number analyzed (Participants) | 16 | 13
  Change at Day 14: Appetite | 0.9 (3.0) | 0.4 (3.9)
  Change at Day 28: Appetite: number analyzed (Participants) | 7 | 6
  Change at Day 28: Appetite | 0.4 (3.1) | -2.0 (2.3)
  Change at Day 7: Well-being: number analyzed (Participants) | 18 | 20
  Change at Day 7: Well-being | -0.8 (2.6) | -0.4 (3.1)
  Change at Day 14: Well-being: number analyzed (Participants) | 16 | 13
  Change at Day 14: Well-being | 0.4 (2.5) | -0.5 (4.3)
  Change at Day 28: Well-being: number analyzed (Participants) | 7 | 6
  Change at Day 28: Well-being | 0.4 (2.4) | -2.3 (2.9)
  Change at Day 7: Shortness of breath: number analyzed (Participants) | 18 | 20
  Change at Day 7: Shortness of breath | -0.1 (2.3) | 0.7 (2.6)
  Change at Day 14: Shortness of breath: number analyzed (Participants) | 16 | 13
  Change at Day 14: Shortness of breath | 0.6 (3.4) | 0.7 (2.9)
  Change at Day 28: Shortness of breath: number analyzed (Participants) | 7 | 6
  Change at Day 28: Shortness of breath | -0.4 (2.0) | -0.2 (3.8)

5. Secondary Outcome: Mean Change From Baseline in Performing General Activity (Karnofsky Performance Status [KPS]); ITT Population
Description: The KPS allows patients to be classified as to their functional impairment and was used to assess general activity. KPS scores range from 0 (dead) to 100 (normal/no disease) and are classified as 0-40 = unable to care for self; 50-70 = unable to work; 80-100 = able to work. The lower the KPS score, the worse the survival for most serious illnesses. Scores were recorded on the patient's medical file at each study visit (Days 1, 7, 14 and 28).
  Mean change from baseline of KPS score at Days 7, 14 and 28 is presented for the ITT population (all randomised patients); a negative change indicates a worsening condition.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Scores on a scale
  Change at Day 7: number analyzed (Participants) | 18 | 19
  Change at Day 7 | -2.8 (12.3) | -3.7 (6.8)
  Change at Day 14: number analyzed (Participants) | 16 | 13
  Change at Day 14 | -5.6 (11.5) | -5.4 (12.7)
  Change at Day 28: number analyzed (Participants) | 8 | 7
  Change at Day 28 | -5.0 (16.0) | -7.1 (20.6)

6. Secondary Outcome: Mean Change From Baseline in Daily Intensity of Abdominal Pain Score (Visual Analogue Scale [VAS]); ITT Population
Description: Abdominal pain was assessed using the VAS numeric pain distress scale which is a 100-millimetre (10-centimetre) scoring scale on which patients mark their perceived level of pain. Scores range from 0 to 100 where 0=no pain and 100=unbearable pain. Higher scores indicate a worse outcome. Scores were recorded on the Patient Diary daily until the end of study (Day 28), by the patient or filled in by the nurse/caregiver in case of patient's physical inability.
  Mean change from baseline of VAS for abdominal pain at Days 7, 14 and 28 is presented for the ITT population; a positive change indicates a worsening condition.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Scores on a scale
  Change at Day 7: number analyzed (Participants) | 19 | 19
  Change at Day 7 | -22.0 (32.5) | -9.6 (30.8)
  Change at Day 14: number analyzed (Participants) | 16 | 14
  Change at Day 14 | -15.6 (34.9) | -27.7 (28.8)
  Change at Day 28: number analyzed (Participants) | 7 | 7
  Change at Day 28 | -32.0 (31.5) | -17.0 (34.9)

7. Secondary Outcome: Number of Patients Experiencing ≤ 2 Vomiting Episodes/Day During at Least 3 Consecutive Days, in Patients Without NGT
Description: Vomiting episodes and NGT presence were recorded on the Patient Diary daily until the end of study (Day 28), by the patient or filled in by the nurse/caregiver in case of patient's physical inability. Number of patients experiencing ≤ 2 vomiting episodes/day during at least 3 consecutive days, in patients without NGT, is presented.
Time Frame: From Baseline (Day 1, before randomisation) to Days 7, 14 and 28.
Population: Patients without NGT were defined as patients without the insertion of NGT for the whole study period. Only patients in the ITT population without NGT and with data available for analysis at each time point are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 6 | 8
Participants
  From Day 1 to Day 7 | 5 | 4
  From Day 1 to Day 14: number analyzed (Participants) | 5 | 7
  From Day 1 to Day 14 | 4 | 4
  From Day 1 to Day 28: number analyzed (Participants) | 5 | 7
  From Day 1 to Day 28 | 4 | 4

8. Secondary Outcome: Mean Daily NGT Secretion Volume, in Patients With a NGT
Description: NGT presence and related secretion volume were recorded on the Patient Diary daily until the end of study (Day 28), by the patient or filled in by the nurse/caregiver in case of patient's physical inability. Mean daily secretion volumes, in patients with NGT, is presented.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: Only patients with NGT and with data available for analysis at each time point are presented.
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 10 | 7
millilitres
  Baseline: number analyzed (Participants) | 1 | 2
  Baseline | 200.0 (NA) — Not calculable as only 1 patient had data available for analysis at this time point. | 700.0 (141.4)
  Day 7: number analyzed (Participants) | 4 | 2
  Day 7 | 4875.0 (4023.6) | 1025.0 (813.2)
  Day 14: number analyzed (Participants) | 2 | 6
  Day 14 | 12675.0 (2863.8) | 7090.8 (2433.9)
  Day 28 | 27501.0 (27081.8) | 18301.4 (11657.9)

9. Secondary Outcome: Mean Change From Baseline in Number of Daily Vomiting Episodes; ITT Population
Description: Vomiting episodes were recorded on the Patient Diary daily until the end of study (Day 28), by the patient or filled in by the nurse/caregiver in case of patient's physical inability. Mean change from baseline in number of daily vomiting episodes is presented for the ITT population.
Time Frame: Baseline (Day 1, before randomisation) and Days 7, 14 and 28.
Population: The ITT population included all randomised patients. Only patients with data available at each time point are presented.
Measure: Mean (Standard Deviation); unit: Episodes (daily)
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Episodes (daily)
  Change at Day 7: number analyzed (Participants) | 21 | 20
  Change at Day 7 | 5.7 (6.2) | 6.0 (9.9)
  Change at Day 14: number analyzed (Participants) | 21 | 20
  Change at Day 14 | 10.6 (12.7) | 10.4 (15.8)
  Change at Day 28: number analyzed (Participants) | 21 | 20
  Change at Day 28 | 16.5 (19.9) | 14.1 (20.2)

10. Secondary Outcome: Assessment of Passage of Stools; ITT Population
Description: Passage of stools assessments (Yes/No) were recorded on the Patient Diary daily until the end of study (Day 28), by the patient or filled in by the nurse/caregiver in case of patient's physical inability.
Time Frame: From Baseline (Day 1, before randomisation) to Day 28.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
Number analyzed (Participants) | 21 | 22
Participants
  Day 1: Yes | 2 | 2
  Day 1: No | 19 | 20
  Day 2: number analyzed (Participants) | 19 | 19
  Day 2: Yes | 6 | 3
  Day 2: No | 13 | 16
  Day 3: number analyzed (Participants) | 19 | 20
  Day 3: Yes | 4 | 3
  Day 3: No | 15 | 17
  Day 4: number analyzed (Participants) | 19 | 20
  Day 4: Yes | 4 | 2
  Day 4: No | 15 | 18
  Day 5: number analyzed (Participants) | 19 | 20
  Day 5: Yes | 6 | 3
  Day 5: No | 13 | 17
  Day 6: number analyzed (Participants) | 19 | 19
  Day 6: Yes | 4 | 2
  Day 6: No | 15 | 17
  Day 7: number analyzed (Participants) | 19 | 19
  Day 7: Yes | 3 | 3
  Day 7: No | 16 | 16
  Day 8: number analyzed (Participants) | 18 | 20
  Day 8: Yes | 6 | 3
  Day 8: No | 12 | 17
  Day 9: number analyzed (Participants) | 17 | 19
  Day 9: Yes | 4 | 5
  Day 9: No | 13 | 14
  Day 10: number analyzed (Participants) | 16 | 16
  Day 10: Yes | 3 | 1
  Day 10: No | 13 | 15
  Day 11: number analyzed (Participants) | 15 | 15
  Day 11: Yes | 5 | 1
  Day 11: No | 10 | 14
  Day 12: number analyzed (Participants) | 15 | 12
  Day 12: Yes | 4 | 1
  Day 12: No | 11 | 11
  Day 13: number analyzed (Participants) | 15 | 14
  Day 13: Yes | 3 | 1
  Day 13: No | 12 | 13
  Day 14: number analyzed (Participants) | 15 | 15
  Day 14: Yes | 5 | 1
  Day 14: No | 10 | 14
  Day 15: number analyzed (Participants) | 14 | 12
  Day 15: Yes | 2 | 2
  Day 15: No | 12 | 10
  Day 16: number analyzed (Participants) | 14 | 11
  Day 16: Yes | 3 | 2
  Day 16: No | 11 | 9
  Day 17: number analyzed (Participants) | 14 | 12
  Day 17: Yes | 2 | 3
  Day 17: No | 12 | 9
  Day 18: number analyzed (Participants) | 14 | 10
  Day 18: Yes | 3 | 2
  Day 18: No | 11 | 8
  Day 19: number analyzed (Participants) | 11 | 10
  Day 19: Yes | 3 | 2
  Day 19: No | 8 | 8
  Day 20: number analyzed (Participants) | 11 | 10
  Day 20: Yes | 2 | 2
  Day 20: No | 9 | 8
  Day 21: number analyzed (Participants) | 11 | 9
  Day 21: Yes | 2 | 2
  Day 21: No | 9 | 7
  Day 22: number analyzed (Participants) | 11 | 8
  Day 22: Yes | 2 | 2
  Day 22: No | 9 | 6
  Day 23: number analyzed (Participants) | 10 | 7
  Day 23: Yes | 3 | 2
  Day 23: No | 7 | 5
  Day 24: number analyzed (Participants) | 10 | 8
  Day 24: Yes | 3 | 2
  Day 24: No | 7 | 6
  Day 25: number analyzed (Participants) | 9 | 7
  Day 25: Yes | 2 | 2
  Day 25: No | 7 | 5
  Day 26: number analyzed (Participants) | 8 | 8
  Day 26: Yes | 2 | 2
  Day 26: No | 6 | 6
  Day 27: number analyzed (Participants) | 8 | 6
  Day 27: Yes | 1 | 2
  Day 27: No | 7 | 4
  Day 28: number analyzed (Participants) | 7 | 7
  Day 28: Yes | 3 | 2
  Day 28: No | 4 | 5

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) until end of study (Day 28).
Description: Treatment emergent adverse events are reported for the safety population which included all patients who received at least one dose of study therapy.
Arm/Group | Standard Care | Standard Care + Lanreotide Autogel
All-Cause Mortality (participants affected / at risk) | 2/21 | 2/22
Serious Adverse Events (participants affected / at risk) | 2/21 | 2/22
Other Adverse Events (participants affected / at risk) | 5/21 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=21) | Standard Care + Lanreotide Autogel (N=22)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=21) | Standard Care + Lanreotide Autogel (N=22)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated early due to insufficient recruitment. As a consequence, the results of the analyses should be interpreted cautiously and no conclusions should be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results are owned by the Sponsor and data communication collected in a center by the investigator is allowed only after publication of aggregate results of the study by the Sponsor. If an investigator intends to communicate data, the Sponsor must be informed and should review the manuscript/publication before its submission. The investigator should accept any Sponsor comments provided they are not in contrast to the reliability of data, with rights, with the safety and well-being of patients.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02365584/SAP_000.pdf
  • Study Protocol (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02365584/Prot_001.pdf